CLINICAL TRIAL: NCT06460636
Title: Combined Effects of Progressive Relaxation Exercises and Aquatic Therapy on Clinical Symptoms, Physical Function and Quality of Life in Patients With Fibromyalgia.
Brief Title: Combined Effects of Progressive Relaxation Exercises and Aquatic Therapy in Fibromyalgia.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0585
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Fibromyalgia
Keywords: Aquatic Therapy; fibromyalgia; physical function; progressive relaxation exercises; quality of life
MeSH Terms: conditions — Fibromyalgia | interventions — Aquatic Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive muscle relaxation therapy + Aquatic therapy (Experimental): Participants in group B will receive progressive muscle relaxation therapy and aquatic therapy. Sessions will be conducted twice a week for 8 weeks and duration will be 30 minutes. 16 sessions overall
  Interventions: Other: progressive muscle relaxation therapy; Other: aquatic therapy
- Progressive muscle relaxation therapy (Active Comparator): Participants in group A will receive progressive muscle relaxation therapy. Sessions will be conducted twice a week for 8 weeks and duration will be 30 minutes. 16 sessions overall
  Interventions: Other: progressive muscle relaxation therapy

INTERVENTIONS:
Other: progressive muscle relaxation therapy — Participants will undergo progressive relaxation exercises, including muscle tension and release with deep breathing, held for 5 seconds each. Sessions will be conducted twice a week for 8 weeks and duration will be 30 minutes. 16 sessions overall
Other: aquatic therapy — participants will receive aquatic therapy. Sessions will be conducted twice a week for 8 weeks and duration will be 30 minutes. 16 sessions overall.
  Arms: Progressive muscle relaxation therapy + Aquatic therapy

SUMMARY:
Fibromyalgia, a chronic pain disorder, presents a significant challenge in healthcare due to its widespread musculoskeletal pain, tenderness, and a spectrum of associated symptoms. This condition profoundly affects patients' physical functions and quality of life, necessitating effective therapeutic interventions. In this study progressive relaxation technique and aquatic therapy with progressive relaxation technique will be used. In aquatic therapy the buoyancy and water resistance play an important role in pain management. This research project aims to explore the efficacy of a novel therapeutic approach by combining progressive relaxation exercises with aquatic therapy.

This will be a randomized controlled trial in which non-probability convenience sampling technique will be used. Sample size will be 54 and this study will be conducted in city hospital, Rahim Yar khan. The study duration will be 7 months participants will be divided into 2 groups (27 in each group). The data will be assessed pre values and post values after 8 week of treatment with the help of visual analog scale for pain, fibromyalgia impact questionnaire, berg balance scale, fatigue severity scale and timed up and go. Data will be analyzed with SPSS version 25.

DETAILED DESCRIPTION:
Fibromyalgia, a chronic pain disorder, presents a significant challenge in healthcare due to its widespread musculoskeletal pain, tenderness, and a spectrum of associated symptoms. This condition profoundly affects patients' physical functions and quality of life, necessitating effective therapeutic interventions. Current treatments primarily focus on symptom management, as there is no known cure for fibromyalgia. There are different interventions used to treat fibromyalgia for example aerobic exercises, resistance exercises, myofascial massage, lymphatic massage. In this study progressive relaxation technique and aquatic therapy with progressive relaxation technique will be used. In aquatic therapy the buoyancy and water resistance play an important role in pain management. This research project aims to explore the efficacy of a novel therapeutic approach by combining progressive relaxation exercises with aquatic therapy.

This will be a randomized controlled trial in which non-probability convenience sampling technique will be used. Sample size will be 54 and this study will be conducted in city hospital, Rahim Yar khan. The study duration will be 7 months participants will be divided into 2 groups (27 in each group). The data will be assessed pre values and post values after 8 week of treatment with the help of visual analog scale for pain, fibromyalgia impact questionnaire for quality of life, berg balance scale, fatigue severity scale for clinical symptoms of fibromyalgia and timed up and go will be used to assess the physical functioning in patients. Data will be analyzed with SPSS version 25.

Keywords: Aquatic Therapy, Fibromyalgia, Physical Function, Progressive Relaxation Exercises, Quality of Life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with age of 20-39 years will be included in this study
2. Married females
3. Only female patients will be included in this study.
4. Diagnosis of fibromyalgia according to established criteria of the American College of Rheumatology (I-e widespread pain index (WPI) ≥7 and symptom severity (SS) scale score ≥5 or WPI 3 - 6 and SS scale score ≥9. Symptoms present at least 3 months(2).
5. Patients having Pain in 11 of 18 tender points will be included.

Exclusion Criteria:

1. Patients with Severe cardiovascular issues will be excluded.
2. Patients with recent injuries or surgeries within the last 6 months will be excluded.
3. Patients with untreated psychiatric disorders will be excluded.

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female (fibromyalgia)
Enrollment: 54 (Estimated)
Dates: Start 2023-12-10 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 8 weeks
  The VAS is a simple and commonly used tool in pain assessment. It consists of a 10 cm line, with endpoints defining extreme limits such as 'no pain' and 'worst imaginable pain.' Participants mark on the line the point that they feel represents their perception of their current state of pain(19). High reliability ICC=0.99(95%CI 0.989 to 0.992). Scoring: The score is determined by measuring the distance from the 'no pain' end of the line to the point that the patient marks.
Fibromyalgia Impact Questionnaire (FIQ) | 8 weeks
  Purpose: To assess the impact of fibromyalgia on daily living. COMBINED EFFECTS OF PROGRESSIVE RELAXATION TECHNIQUE AND AQUATIC THERAPY PATIENTS WITH FIBROMYALGIA 10 Description: The FIQ is a specific questionnaire designed for fibromyalgia patients. It covers aspects such as physical functioning, work status, depression, anxiety, sleep, pain, stiffness, fatigue, and well-being(20). Reliability 0.56 of pain score to 0.95 for physical function.
  Scoring: It consists of 10 items, each scored on a scale, providing a total score that reflects the overall impact of fibromyalgia on the patient.
Berg Scale Test | 8 weeks
  The Berg Balance Scale is a testing tool with high validity and reliability used to measure balance. Balance gives an individual the ability to achieve physical movement and further carry out the activities of daily living. Balance can be classified as either static or dynamic. Fibromyalgia is a common chronic pain condition that exerts a considerable impact on a patient's daily activities and quality of life(
Fatigue Severity Scale | 8 weeks
  The Fatigue Severity Scale (FSS) is a 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle. A self-report scale of nine items about fatigue, its severity and how it affects certain activities. Answers are scored on a seven-point scale where 1 = strongly disagree and 7 = strongly agree. This means the minimum score possible is nine and the highest is 63. The higher the score, the more severe the fatigue is and the more it affects the person's activities. Correlates with depressive symptoms (Beck Depression Inventory) and quality of life(
timed up and go test | 8 weeks
  Mobility is assessed based on time to complete the test: < 10 seconds = normal. < 20 seconds = good mobility; can walk outside alone; does not require a walking aid. < 30 seconds = walking and balance problems; cannot walk outside alone; requires walking aid

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha Arshad, M.phill, Principal Investigator — Riphah International University
Locations (1):
- City Hospital, Rahim Yar Khan, Rahim Yar Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ma J, Zhang T, Li X, Chen X, Zhao Q. Effects of aquatic physical therapy on clinical symptoms, physical function, and quality of life in patients with fibromyalgia: A systematic review and meta-analysis. Physiother Theory Pract. 2024 Feb;40(2):205-223. doi: 10.1080/09593985.2022.2119906. Epub 2022 Sep 4. PMID 36062580
- [Background] Kiyak S, Kocoglu-Tanyer D. Effectiveness of progressive muscle relaxation and laughter therapy on mental health and treatment outcomes in women undergoing in vitro fertilization: A randomized controlled trial. Res Nurs Health. 2021 Dec;44(6):945-956. doi: 10.1002/nur.22187. Epub 2021 Oct 3. PMID 34605040
- [Background] Viveiro LAP, Gomes GCV, Bacha JMR, Carvas Junior N, Kallas ME, Reis M, Jacob Filho W, Pompeu JE. Reliability, Validity, and Ability to Identity Fall Status of the Berg Balance Scale, Balance Evaluation Systems Test (BESTest), Mini-BESTest, and Brief-BESTest in Older Adults Who Live in Nursing Homes. J Geriatr Phys Ther. 2019 Oct/Dec;42(4):E45-E54. doi: 10.1519/JPT.0000000000000215. PMID 30407272
- [Background] Naik H, Shao S, Tran KC, Wong AW, Russell JA, Khor E, Nacul L, McKay RJ, Carlsten C, Ryerson CJ, Levin A. Evaluating fatigue in patients recovering from COVID-19: validation of the fatigue severity scale and single item screening questions. Health Qual Life Outcomes. 2022 Dec 27;20(1):170. doi: 10.1186/s12955-022-02082-x. PMID 36575437